CLINICAL TRIAL: NCT01033266
Title: Effect of Continuous Positive Airway Pressure (CPAP) and Cardiopulmonary Exercise Testing(CPET) in Patient With Obstructive Sleep Apnea (OSA) and Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: Effect of Nasal CPAP on Cardiopulmonary Exercise Testing in Patients With Overlap Syndrome
Status: Completed | Type: Observational
Sponsor: University of Oklahoma (Other)
Responsible Party: Sponsor
Other Study IDs: 14587/2895
Record Dates: First submitted 2009-12-15; First posted 2009-12-16 (Estimated); Last update posted 2020-04-14 (Actual); Status verified 2020-04

CONDITIONS: Obstructive Sleep Apnea; Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Sleep Apnea, Obstructive; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- CPET CPAP
  Interventions: Diagnostic Test: CPET

INTERVENTIONS:
Diagnostic Test: CPET — CPET will be done on patients with overlap syndrome before and after clinical CPAP treatment.

SUMMARY:
Nasal CPAP will improve cardiopulmonary exercise test (CPET) performance in patients with overlap syndrome(COPD and OSA). Nasal CPAP is proven to improve cardiopulmonary exercise testing in patients with OSA. The investigators hypothesis is that patients with overlap syndrome will have a greater improvement in their cardiopulmonary exercise testing besides a possible improvement in their lung function test and airway resistance.

DETAILED DESCRIPTION:
Patients presenting to the Oklahoma City VA sleep clinic with obstructive sleep apnea syndrome and a desire to initiate CPAP treatment will be included if they have overlap syndrome. Patients will undergo a spirometry and CPET before being started on CPAP as part of standard clinical care. The CPET will be repeated after 8-12 weeks of CPAP use. Patients will be excluded if they have any contraindication to mild exercise or they cannot perform an exercise test due to limited mobility.

ELIGIBILITY:
Inclusion Criteria:

* Obstructive sleep apnea (OSA)
* COPD

Exclusion Criteria:

* Inability to perform exercise test due to musculoskeletal limitation
* Cardiac condition preventing patient from mild exercise
* Continuous oxygen supplement

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with OSA and COPD will perform CPET before and after use of CPAP.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2009-02-01 (Actual); Primary Completion 2014-02-28 (Actual); Study Completion 2014-02-28 (Actual)

PRIMARY OUTCOMES:
Efficacy of nasal CPAP on CPET performance in patients with overlap syndrome | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Gary Kinasewitz, MD, Principal Investigator — University of Oklahoma; Houssein Youness, MD, Principal Investigator — University of Oklahoma
Locations (2):
- United States (2):
  - OU Medical Center, Oklahoma City, Oklahoma
  - VA Medical Center, Oklahoma City, Oklahoma